CLINICAL TRIAL: NCT00752271
Title: Inflammatory and Biomechanical Contributors to Arthritis Development Following Arthroscopic Meniscectomy
Brief Title: AMS Study: Inflammatory and Biomechanical Contributors to Arthritis Development Following Arthroscopic Meniscectomy
Status: Terminated | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Shari M. Ling, MD, National Institute on Aging
Other Study IDs: AG0105
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-12

CONDITIONS: Osteoarthritis
Keywords: Arthroscopic
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 24 adults with meniscal damage for which arthroscopy is clinically indicated
- 2: 8 adults who have already undergone meniscal resection to serve as positive controls

SUMMARY:
The purpose of this study is to examine the relationship between muscle activation and heart rate on joint generalized inflammation and arthritis development.

DETAILED DESCRIPTION:
This study will test the hypothesis that knee trauma (as exemplified by the arthroscopy procedure) causes inflammation that alters muscle activation patterns locally and also disrupts the balance between parasympathetic-sympathetic reflexes. It is hypothesized that these factors contribute to development and progression of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 or older
* Potential candidate for knee arthroscopy for medial
* Meniscal tear confirmed on MRI
* Prior meniscal resection at least 1 year prior with a persistent knee effusion
* Body mass index between 25-35 kg/m2

Exclusion Criteria:

* Knee injury in the 1 month before the initial study evaluation
* Knee surgery within 1 year before the initial study evaluation
* Pace-maker or defibrillator, 2nd or 3rd degree heart block, or other abnormal rhythms
* Current diagnosis of diabetes mellitus, a fasting glucose>100mg/dl or >140 mg/dl 2 hour after a glucose challenge
* Current diagnosis of an inflammatory condition (e.g. rheumatoid arthritis, gout, etc)
* Untreated thyroid disease
* Morbid obesity (body mass index >35)
* Neuropathy or nerve damage
* Stroke or transient-ischemic attacks (mini-stroke)
* Recent diagnosis of congestive heart failure or heart attack
* Use of prednisone or chemotherapy, steroid or other joint or ant-inflammatory agents in the past 3 months
* Current use of medications that influence heart rate
* Cognitive impairment that limits your ability to provide informed consent
* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Orthopedic and arthritis clinics in the Baltimore/Washington DC area
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shari M. Ling, MD, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- NIA Clinical Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Handel TM, Johnson Z, Crown SE, Lau EK, Proudfoot AE. Regulation of protein function by glycosaminoglycans--as exemplified by chemokines. Annu Rev Biochem. 2005;74:385-410. doi: 10.1146/annurev.biochem.72.121801.161747. PMID 15952892
- [Background] Roos EM. Joint injury causes knee osteoarthritis in young adults. Curr Opin Rheumatol. 2005 Mar;17(2):195-200. doi: 10.1097/01.bor.0000151406.64393.00. PMID 15711235
- [Background] Saeed RW, Varma S, Peng-Nemeroff T, Sherry B, Balakhaneh D, Huston J, Tracey KJ, Al-Abed Y, Metz CN. Cholinergic stimulation blocks endothelial cell activation and leukocyte recruitment during inflammation. J Exp Med. 2005 Apr 4;201(7):1113-23. doi: 10.1084/jem.20040463. PMID 15809354